CLINICAL TRIAL: NCT04442542
Title: Method JaPer. A New Strategy to Improve Inspirational Capacity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Tolteca (Other)
Responsible Party: Principal Investigator, Javier Eliecer Pereira Rodriguez, Physiotherapist, specialist in cardiopulmonary rehabilitation, master in palliative care, University Tolteca
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: JEPereiraRodriguez
Record Dates: First submitted 2020-06-18; First posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Inspiratory Capacity
Keywords: Inspiratory Capacity; physiotherapy; pulmonar rehabilitation
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: 850 hospitalized patients, who, after the exclusion criteria, 708 hospitalized patients with different diseases (mainly cancer, heart failure, COPD, postoperative gastrointestinal, fractures, pneumonia, high blood pressure, diabetes mellitus) finally began the investigation and organized into 2 groups. The present one was distributed with a basic probability sampling using a table of random numbers, the order of which was randomized through the Microsoft Excel 16.0 program, with the experimental group being 337 participants (Respiratory exercises plus new method of intervention with respiratory incentive - JaPer Method -) and the control group with 371 (Respiratory exercises plus conventional use of the respiratory incentive).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Respiratory exercises plus method JaPer (Experimental): Respiratory exercises plus the new intervention protocol with an inspirometer (JaPer Method)
  Interventions: Other: Respiratory muscle training 1 (Experimental Group)
- Protocol of use of inspirometer in a conventional way (Active Comparator): Respiratory exercises plus conventional use of the inspirometer.
  Interventions: Other: Respiratory muscle training 2 (Control Group)

INTERVENTIONS:
Other: Respiratory muscle training 1 (Experimental Group) — The participant must perform a series of exercises that will be the same for the two groups in this investigation. In addition to the exercises, this group will use the incentive inspirometer device with a new method created by the main author called the Method JaPer.
  For the method JaPer, the participant sits and holds the device. Then put the mouthpiece of the inspirometer in the mouth. Be sure to make a good seal on the mouthpiece with your lips. And exhale normally until you run out of air. And after that, inhale slowly as much as possible. This maximum value will be taken as an indicative parameter of its maximum inspiratory capacity and 50 and 80% for 1 set of 10 repetitions at 50% of their maximum value, 2 sets of 10 repetitions at 60% of its maximum capacity and ends with 1 series at 80% of its maximum capacity. It is highlighted that in each series before finishing and without stopping to rest, the participant must do 5 repetitions at 100% maximum capacity
  Other Names: Method JaPer
  Arms: Respiratory exercises plus method JaPer
Other: Respiratory muscle training 2 (Control Group) — Training of respiratory muscles under the protocol of conventional use. Which is that the participant sits and holds the device. Then put the mouthpiece of the inspirometer in the mouth. Be sure to make a good seal on the mouthpiece with your lips. And exhale (exhale) normally until you run out of air. And after that, inhale (inspire) slowly as much as possible. Repeat 10 times and use these indications for 3 sets. In addition, participants must perform the same breathing exercises that are identical for experimental group.
  Arms: Protocol of use of inspirometer in a conventional way

SUMMARY:
Different diseases worldwide have repercussions at the level of multiple systems; but without a doubt a higher prevalence in the cardiopulmonary system. When a patient is hospitalized, he enters a continuous and often prolonged rest stay. Wherein, this physical inactivity plus its base pathology negatively impact its lung capacity. And low lung capacity has been shown to increase the risk of mortality, hospital stay, and complications. That said, the use of the device known as the "incentive inspirometer" is important, which to some extent there is no standardization of its use or applicability in a structured and planned manner. For this reason, the Japer method emerges as an idea; which, pretending through an exercise prescription through the incentive inspirometer according to 50% to 80% of the maximum inspiring capacity of the patient, improves their inspiring capacity. Having said this, the general objective was to analyze the effects of the JaPer method to improve lung capacity versus the traditional use of an inspirometer in hospitalized patients.

DETAILED DESCRIPTION:
In 1974 the Respiratory Rehabilitation (RR) Committee of the American College of Chest Physicians defined RR as an art. It took almost 20 more years for another group of experts to describe it as a service. Moving forward in our reasoning, it is important to remember that all physical activity produces an increase in metabolic energy expenditure, as a result of body movement carried out in a specific period of time. The current literature through various organizations has been oriented to promote activities that arouse interest in generating movement and thus obtain benefits in improving health and quality of life. The respiratory physiotherapy techniques are basically divided into 2 types: facilitating techniques for expectoration and respiratory exercises. The former are indicated in hypersecretory processes, in alterations in the properties of mucus, ciliary dysfunction and alterations in the cough mechanism, to keep the airway free of secretions. The second is focused on improving a respiratory pattern, a respiratory reeducation, strengthening of respiratory muscles, preventing and / or reducing dyspnea and fatigue through the use of the inspirometer, respiratory exercises and specific techniques. In addition, it helps to decrease the hospital stay. Which, when prolonged, generates negative effects on the health system, such as: increased costs, poor accessibility to hospitalization services, saturation of emergencies and risks of adverse events. Plus all the negative effects it can generate in a hospitalized patient.

Different diseases worldwide have repercussions at the level of multiple systems; but without a doubt a higher prevalence in the cardiopulmonary system. When a patient is hospitalized, he enters a continuous and often prolonged rest stay. Wherein, this physical inactivity plus its base pathology negatively impact its lung capacity. And low lung capacity has been shown to increase the risk of mortality, hospital stay, and complications. That said, the use of the device known as the "incentive inspirometer" is important, which to some extent there is no standardization of its use or applicability in a structured and planned manner. For this reason, the Japer method emerges as an idea; which, pretending through an exercise prescription through the incentive inspirometer according to 50% to 80% of the maximum inspiring capacity of the patient, improves their inspiring capacity. Having said this, the general objective was to analyze the effects of the JaPer method to improve lung capacity versus the traditional use of an inspirometer in hospitalized patients.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients cardiopulmonary pathologies
* Over 18 years of age
* Patients who sign informed consent
* Possibility of performing your training for 1 month
* Participants than will can to go everyday for intervention.
* Participants do not have any inconvenience when doing the questionnaires, tests and measures that the investigation demands.

Exclusion Criteria:

* Participants who had severe pain in the lower or upper limbs.
* Unstable angina.
* Heart rate >120 bpm (beats per minute) at rest.
* Systolic blood pressure >190 mmHg.
* Diastolic blood pressure >120 mmHg.
* Participants who had a positive contraindication make exercise were not admitted in the study.
* Participants to show hemodynamic instability without improving during any test or during the intervention process.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 708 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Maximum inspiratory volume (ml) | 2 week
  It will be determined by using the inspirometer whose values are from 0ml to 5,000ml. This pre and post intervention value will be determined
Changes in the levels of Fatigue after intervention | 2 week
  Fatigue was assessed using the FACT-Fatigue Scale Scale (Fatigue Scale of the Functional Evaluation of Cancer Therapy), which is an inventory of 13 items that assesses the severity of cancer-associated fatigue (FAC) in the last week. with a scale of 0 to 4 and that with higher scores reflect a lower FAC.
Changes in the Dyspnoea a after intervention | 2 week
  Dyspnea is a respiratory difficulty that usually translates into shortness of breath. Dyspnea can be determined using the original Borg scale (Score from 0 to 20) or modified (Score from 0 to 10), in which the higher the number indicated by the participant, the higher the degree of dyspnea.
Changes in the levels of Quality of life after intervention: EORTC QLQ-C30 | 2 week
  For the quality of life, it is necessary to use the questionnaire called EORTC QLQ-C30 (Version 3), which has 30 questions, where each question will go with a score of 1 to 4 and the higher the final result the better the quality of life. participant's life.
Changes in the Estimated maximum oxygen volume after 15 training sessions (ml/kg/min) | 2 week
  It is the maximum amount of oxygen that the body can absorb, transport and consume in a given time, is the blood that our body can transport and metabolize. To determine the Vo2 values, the 6-minute walking test is used and to determine the result of the test, formulas are used according to the meters traveled, age, sex, height and weight of the participant. The larger the meters traveled, the greater the vo2.
Changes in the unit of measurement of the metabolic index (METs) after 15 training sessions (ml/kg/min) | 2 week
  It is the unit of measurement of the metabolic index (amount of energy consumed by an individual in a resting situation). To determine the METs values, the 6-minute walking test is used and to determine the result of the test, formulas are used according to the meters traveled, age, sex, height and weight of the participant. The larger the meters traveled, the greater the METs.
Changes in the Distance traveled after 15 training sessions (m) | 2 week
  Distance traveled in this of 6 minute walk test. The larger the meters traveled, this will indicate better Vo2, METs and aerobic and physical capacity in the participant.

SECONDARY OUTCOMES:
Changes of the maximum heart rate in a effort test after 15 training sessions | 2 week
  It is the maximum capacity that the heart has to contract and we determine it by means of an effort test. The Maximum heart rate can be determined by formula or in a effort test (In the present investigation) which consists in mounting the participant in an endless band with an inclination and speed determined according to the protocol for said test. The test is stopped when the participant. indicates that it can not be more or there are electrocardiographic alterations that indicate that it is the participant's maximum.
Changes in the Body weight after 15 training sessions (Kg) | 2 week
  How much body weight (kg) pre and post intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Tolteca - Puebla, Puebla City, Mexico

IPD SHARING:
Plan to Share IPD: No
We don ́t have any plan because The research will be carried out directly among the researchers of our center. However, it is highlighted that we will make our results available to other researchers so that they can carry out future research that supports our results and compares with other types of populations.